CLINICAL TRIAL: NCT06231329
Title: The Role of Ultrasound Elastography in the Diagnosis of Testicular Tumors
Brief Title: Role of Elastography in Diagnosis of Testicular Tumors
Status: Not yet recruiting | Type: Observational
Sponsor: Ali Mohamed Alaa El-din (Other)
Responsible Party: Sponsor-Investigator, Ali Mohamed Alaa El-din, Resident at radiology department, Assiut University
Organization: Assiut University (Other)
Other Study IDs: elastography testicular tumors
Record Dates: First submitted 2024-01-20; First posted 2024-01-30 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Testicular Cancer
MeSH Terms: conditions — Testicular Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: ultrasound elastography — examining patient's testis with ultrasound elastography technique and collect data and results

SUMMARY:
The aim of study is to differentiate between testicular tumors by their elastographic criteria (Stiffness [hard to soft] , Shape under compression , etc.) using ultrasound elastography techniques (shear wave/strain elastography) on suspected testicle that showed specific lesion on normal ultrasound examination.

DETAILED DESCRIPTION:
Technique:

Using a linear ultrasound probe supporting elastography techniques, either :

Strain Elastography (SE) SE measures tissue stiffness by applying external tissue pressure [3]. Tissue dimensions change due to the applied pressure; this deformation is termed strain. Stiffer lesions deform less, and have correspondingly lower strain and higher Young's modulus.

In strain imaging, tissue displacement is calculated by processing radiofrequency (RF) datasets obtained before and after compression [4]. Translucent colored elastograms (strain images) can be superimposed on B-mode images to provide complementary anatomic information. It is common to display the strain map as colored pixels on a red/blue scale or gray scale [5].

Or Shear wave elastography (SWE) Shear wave elastography differs from strain elastography, as it is a quantitative method of assessing tissue elasticity by measuring the speed of acoustic radiation force impulse-induced shear waves traveling in the tissue of interest.

The compressive acoustic waves used for conventional B-mode image generation travel at high speeds through soft tissue (1450-1550 m/s). By contrast, mechanical shear waves used for shear wave elastography travel relatively slowly (1-10 m/s). Shear wave propagation velocity depends on tissue stiffness [2, 4].

Data collection:

Data will be recorded as excel spreadsheet and statistical analysis using SPSS software version 22

Computer software: SPSS version 22 statistical software.

Statistical tests: T-test.

ELIGIBILITY:
Inclusion Criteria:

* i. Age : (15-65 years).
* ii. Patient with history of testicular pain or discomfort or even without clinical symptoms.
* iii. Patient with any predisposing factors as mentioned before in the background.
* iv. Patient with history of cancer of other organs (not testicular tumors).

Exclusion Criteria:

* i. patient refused to be included in the study. ii. infarct correlation with patient history and symptoms is important. iii. Infections as focal orchitis. iv. History of trauma (hematoma exclusion).

Ages: 15 Years to 65 Years | Sex: Male
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: male patients with testicular mass lesion
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
collect data of our elastography examination and acknowledge more information about certain testicular tumors and percentage of malignant and bengin tumors of our specimen using ultrasound machine shear wave mode | baseline
  differentiate between certain types of testicular tumors according to their elastography criteria using ultrasound machine shear wave mode according to the elasticity of tumor tissue

REFERENCES:
- [Background] Stephenson A, Eggener SE, Bass EB, Chelnick DM, Daneshmand S, Feldman D, Gilligan T, Karam JA, Leibovich B, Liauw SL, Masterson TA, Meeks JJ, Pierorazio PM, Sharma R, Sheinfeld J. Diagnosis and Treatment of Early Stage Testicular Cancer: AUA Guideline. J Urol. 2019 Aug;202(2):272-281. doi: 10.1097/JU.0000000000000318. Epub 2019 Jul 8. PMID 31059667
- [Background] Gilligan T, Lin DW, Aggarwal R, Chism D, Cost N, Derweesh IH, Emamekhoo H, Feldman DR, Geynisman DM, Hancock SL, LaGrange C, Levine EG, Longo T, Lowrance W, McGregor B, Monk P, Picus J, Pierorazio P, Rais-Bahrami S, Saylor P, Sircar K, Smith DC, Tzou K, Vaena D, Vaughn D, Yamoah K, Yamzon J, Johnson-Chilla A, Keller J, Pluchino LA. Testicular Cancer, Version 2.2020, NCCN Clinical Practice Guidelines in Oncology. J Natl Compr Canc Netw. 2019 Dec;17(12):1529-1554. doi: 10.6004/jnccn.2019.0058. PMID 31805523
- [Background] Wood L, Kollmannsberger C, Jewett M, Chung P, Hotte S, O'Malley M, Sweet J, Anson-Cartwright L, Winquist E, North S, Tyldesley S, Sturgeon J, Gospodarowicz M, Segal R, Cheng T, Venner P, Moore M, Albers P, Huddart R, Nichols C, Warde P. Canadian consensus guidelines for the management of testicular germ cell cancer. Can Urol Assoc J. 2010 Apr;4(2):e19-38. doi: 10.5489/cuaj.815. No abstract available. PMID 20368885
- [Background] Kreydin EI, Barrisford GW, Feldman AS, Preston MA. Testicular cancer: what the radiologist needs to know. AJR Am J Roentgenol. 2013 Jun;200(6):1215-25. doi: 10.2214/AJR.12.10319. PMID 23701056
- [Background] Necas M, Muthupalaniappaan M, Barnard C. Ultrasound morphological patterns of testicular tumours, correlation with histopathology. J Med Radiat Sci. 2021 Mar;68(1):21-27. doi: 10.1002/jmrs.426. Epub 2020 Sep 1. PMID 32869524